CLINICAL TRIAL: NCT00441402
Title: Exercise Amenorrhea Stress and Bone Health in Adolescents
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK65995 (completed)
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study investigates the role of energy balance and stress in the regulation of hypothalamic-pituitary-gonadal axis in adolescent girls across the fitness spectrum.

ELIGIBILITY:
Inclusion Criteria:

* healthy adolescent girls not taking any medications

Exclusion Criteria:

* Hormonal preparation or birth control within 12 months prior to enrollment
* Galactorrhea
* Clinical Depression

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Z. Kasa-Vubu, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Kasa-Vubu JZ, Rosenthal A, Murdock EG, Welch KB. Impact of fatness, fitness, and ethnicity on the relationship of nocturnal ghrelin to 24-hour luteinizing hormone concentrations in adolescent girls. J Clin Endocrinol Metab. 2007 Aug;92(8):3246-52. doi: 10.1210/jc.2006-2852. Epub 2007 May 15. PMID 17504901